CLINICAL TRIAL: NCT05641064
Title: Evaluation of Intraoperative Dexmedetomidine Use on Reducing Inflammatory Response Caused by Cardiopulmonary Bypass in Patients Undergoing Surgical Aortic Valve Replacement
Brief Title: Evaluation of Intraoperative Dexmedetomidine Use in Patients Undergoing Surgical Aortic Valve Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Zrinka Safaric Oremus, Principal Investigator, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 78Z11053
Record Dates: First submitted 2022-11-02; First posted 2022-12-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Systemic Inflammatory Response; Aortic Valve Stenosis
Keywords: dexmedetomidine
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Sodium Chloride; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization and study drug preparation by person(s) not involved in patient care, data gathering or outcome evaluation. Group allocation kept in sealed opaque envelope until all data gathered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Saline (Placebo Comparator): Continuous infusion of saline starting after invasive monitoring placement and before initiation of cardiopulmonary bypass (CPB) until the end of surgery
  Interventions: Drug: Placebo
- Dexmedetomidine 0.5 (Experimental): Continuous infusion of dexmedetomidine in dose 0.5 mcg/kg/min starting after invasive monitoring placement and before initiation of cardiopulmonary bypass (CPB) until the end of surgery
  Interventions: Drug: Dexmedetomidine 0.5mcg/kg/h
- Dexmedetomidine 1 (Experimental): Continuous infusion of dexmedetomidine in dose 1 mcg/kg/min starting after invasive monitoring placement and before initiation of cardiopulmonary bypass (CPB) until the end of surgery
  Interventions: Drug: Dexmedetomidine 1 mcg/kg/h

INTERVENTIONS:
Drug: Placebo — Continuous infusion of saline starting after invasive monitoring placement before cardiopulmonary bypass (CPB) initiation up to surgery completion
  Other Names: saline
  Arms: Saline
Drug: Dexmedetomidine 0.5mcg/kg/h — Continuous infusion of dexmedetomidine in 0.5mcg/kg/h dose starting after invasive monitoring placement before cardiopulmonary bypass (CPB) initiation up to surgery completion
  Other Names: dexmedetomidine in 0.5mcg/kg/h dose
  Arms: Dexmedetomidine 0.5
Drug: Dexmedetomidine 1 mcg/kg/h — Continuous infusion of dexmedetomidine in 1mcg/kg/h dose starting after invasive monitoring placement before cardiopulmonary bypass (CPB) initiation up to surgery completion
  Other Names: dexmedetomidine in 1 mcg/kg/h dose
  Arms: Dexmedetomidine 1

SUMMARY:
Aim of this randomized prospective study is to investigate the immunomodulatory effects of dexmedetomidine on outcomes in patients with isolated aortic stenosis after surgical aortic valve replacement.

DETAILED DESCRIPTION:
Study will investigate effects of two different doses of dexmedetomidine on concentrations of tumor necrosis factor-α and interleukin-6, on inflammatory parameters (C reactive protein and procalcitonin) and inflammatory complications, renal function, postoperative delirium, anaesthetic and analgetic consumption and compare it to control group. It should provide a better understanding of dexmedetomidine effect on decrease of inflammatory response in patients undergoing cardiac surgery. Short-term infusion of dexmedetomidine could reduce inflammatory postoperative complications, contribute to improvement of perioperative renal function and occurrence of postoperative delirium, supporting recovery and shortening hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* isolated aortic stenosis adult patients with written consent

Exclusion Criteria:

* BMI <30kg/m2
* 1st, 2nd and 3rd degree AV block
* bradycardia HR<50/min upon arrival to operating theatre
* neurological disorders (Parkinson's disease, Myasthenia gravis, multiple sclerosis, brain tumors in anamnesis)
* recent use of psychoactive drugs
* alcohol and illicit drug addiction
* diabetes type I with complications
* patients who develop hypotension after initiation of dexmedetomidine infusion requiring vasoconstriction therapy
* patients receiving corticosteroids in perioperative period
* patients with known allergy to dexmedetomidine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-09-22 (Actual); Study Completion 2024-09-22 (Actual)

PRIMARY OUTCOMES:
interleukin 6 | 24 hours preoperatively up to 12 hours post CPB
  Concentration of IL-6 24 hours preoperatively (T0), before CPB initiation (T1), 5 hours post CPB (T2) and 12 hours post CPB (T3)
tumor necrosis factor alpha | 24 hours preoperatively up to 12 hours post CPB
  Concentration of TNF-alpha 24 hours preoperatively (T0), before CPB initiation (T1), 5 hours post CPB (T2) and 12 hours post CPB (T3)

SECONDARY OUTCOMES:
Inflammatory marker concentration during hospital stay | From recruitment date up to 30 days postoperatively
  Determination of concentration of CRP and procalcitonin during hospital stay
Infection rate | From recruitment date up to 30 days postoperatively
  Determining incidence of wound infection, pneumonia, urinary infection and sepsis during hospital stay
Renal function - diuresis | From recruitment date up to 10 days postoperatively
  Determining parameters of renal function: Daily 24-hour urine output in ml
Renal function - diuretic consumption | From recruitment date up to 10 days postoperatively
  Determining parameters of renal function: diuretic consumption
Renal function - GFR | From recruitment date up to 10 days postoperatively
  Determining parameters of renal function: glomerular filtration rate
Renal function - creatinine | From recruitment date up to 10 days postoperatively
  Determining parameters of renal function: creatinine concentration
Renal function - urea | From recruitment date up to 10 days postoperatively
  Determining parameters of renal function: urea concentration
Postoperative delirium | From recruitment date up to 30 days postoperatively
  Determining incidence of postoperative delirium using Confusion Assessment Method questionaire
Analgesic and anesthetic consumption | From recruitment date up to 10 days postoperatively
  Determining intraoperative anesthetic consumption (midazolam, sufentanil, propofol and sevoflurane) and postoperative analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Zrinka Safaric Oremus, MD, Principal Investigator — UH Dubrava
Locations (1):
- University hospital Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma Y, Yu XY, Wang Y. Dose-related effects of dexmedetomidine on immunomodulation and mortality to septic shock in rats. World J Emerg Med. 2018;9(1):56-63. doi: 10.5847/wjem.j.1920-8642.2018.01.009. PMID 29290897
- [Background] Bulow NM, Colpo E, Pereira RP, Correa EF, Waczuk EP, Duarte MF, Rocha JB. Dexmedetomidine decreases the inflammatory response to myocardial surgery under mini-cardiopulmonary bypass. Braz J Med Biol Res. 2016;49(4):e4646. doi: 10.1590/1414-431X20154646. Epub 2016 Feb 23. PMID 26909786
- [Background] Lee JM, Han HJ, Choi WK, Yoo S, Baek S, Lee J. Immunomodulatory effects of intraoperative dexmedetomidine on T helper 1, T helper 2, T helper 17 and regulatory T cells cytokine levels and their balance: a prospective, randomised, double-blind, dose-response clinical study. BMC Anesthesiol. 2018 Nov 8;18(1):164. doi: 10.1186/s12871-018-0625-2. PMID 30409131